CLINICAL TRIAL: NCT06448572
Title: EXL01 in Combination With Nivolumab for Advanced NSCLC Refractory to Immunotherapy
Acronym: EXLIBRIS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Exeliom Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRI_2022/0641; 2023-505285-28-01 (EU CTIS Number)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Immunotherapy; microbiota; Lung Cancer bacteria; Faecalibacterium prausnitzii
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXL01 + Nivolumab (Experimental)
  Interventions: Drug: EXL01

INTERVENTIONS:
Drug: EXL01 — 1 capsule / day

SUMMARY:
As treatment options are limited following progression on anti PD-(L)1 and platinum-based chemotherapy, we propose this trial for patients who have failed to respond or have shown intolerance to standard therapies or for whom no appropriate therapies are known to provide clinical benefit. Considering the strong therapeutic rationale of an association between antineoplastic immunotherapy and EXL01 (single-strain of F. prausnitzii, a bacteria which is a dominant member of the healthy gut microbiota), we propose to assess this combination for NSCLC treatment. This is a pilot, Phase I/II, one-arm, monocentric study evaluating the combination of EXL01 with nivolumab treatment for Non-Small Cell Lung Cancer patients.

ELIGIBILITY:
Key inclusion Criteria:

1. Patients (male or female) ≥18 years old.
2. ECOG Performance status (PS) 0-1 (WHO).
3. Histologically or cytologically documented inoperable advanced/metastatic NSCLC. (inoperable stage III not amenable to radiation therapy or surgery, stage IV)
4. No alterations of key driver oncogenes including EGFR (mutations), ALK (fusions), ROS1 (fusions), MET (METex14 mutations), HER2 (exon 20 insertions), RET (fusions), or BRAF (V600E mutations). KRAS mutations are allowed.
5. Must have previously received anti-PD(L)1 agent and platinum-based chemotherapy, either concomitantly or sequentially. Last dose to have been administered more than 15 days prior to first dose of study drug.
6. Must have progressed within 6 months after first dose of anti-PD(L)1 given either alone or in combination with platinum-based chemotherapy.
7. Must have received all validated available standard therapies.
8. Measurable disease according to iRECIST 1.1.
9. Adequate hematological, renal and liver functions within 72 hours before the first dose of study treatment:

   * Absolute Neutrophil Count ≥ 1500/μL
   * Platelets ≥ 100 000/μL
   * Hemoglobin ≥ 9.0 g/dL
   * Creatinine Clearance ≥ 50 mL/min
   * Total Bilirubin ≤ 1.5 x ULN
   * AST and ALT ≤ 2.5 x ULN (≤ 5 x ULN for participants with liver metastasis)

Key exclusion Criteria:

1. Small cell lung cancer or tumors with mixed histology including a SCLC component.
2. Known symptomatic CNS metastases and/or carcinomatous meningitis. Participants with asymptomatic brain metastases (ie, no neurological symptoms and no requirements for corticosteroids > 10mg/d prednisone equivalent) may participate.
3. Diagnosis of immunodeficiency of is receiving systemic treatment with corticosteroids with greater dose than 10 mg prednisone equivalent daily, within 14 days before initiation of the immunotherapy induction. Inhaled, nasal or topic corticosteroids are allowed.
4. Living attenuated vaccine received within the 30 previous days.
5. Has received Fecal Microbiota Transplantation within 3 months prior to Screening.
6. General serious condition such as uncontrolled congestive cardiac failure, uncontrolled cardiac arrythmia, uncontrolled ischemic cardiac disease (unstable angina or history of myocardial infarction within the previous 6 months), history or stroke within the 6 previous months.
7. History of severe immune-mediated toxicity (≥ grade 3) under immunotherapy treatment.
8. History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate (PFS Rate) for the assessment of efficacy, defined as the rate of alive and non-progressive subjects as per iRECIST 1.1 over the study subjects. | At 3 months from the inclusion

SECONDARY OUTCOMES:
Number of Grade ≥ 3 treatment-related AEs, using CTCAE | First 6 weeks of treatment
Progression Free Survival, defined as the time from inclusion to the first documented disease progression or death due to any cause, whichever occurs first. | First 6 weeks of treatment
ORR (Overall Response Rate) as per iRECIST1.1 for the assessment of efficacy, defined as the rate of confirmed Complete Response (CR) or Partial Response (PR) over the study subjects efficacy responses. | First 6 weeks of treatment
Overall Survival, defined as the time from inclusion to the date of death due to any cause | First 6 weeks of treatment
Disease Control Rate, defined as the rate of confirmed Complete Response (CR), or Partial Response (PR), or Stable Disease (SD) over the study subjects efficacy responses | First 6 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No